CLINICAL TRIAL: NCT04337060
Title: Single-injection Ultrasound-guided Erector Spinae Plane Block for Postoperative Analgesia in Patients Undergoing Open Radical Prostatectomy: A Prospective Randomized Sham-controlled Trial
Brief Title: Open Radical Prostatectomy and Erector Spinae Plane Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BURHAN DOST (Other)
Collaborators: Ondokuz Mayıs University (Other)
Responsible Party: Sponsor-Investigator, BURHAN DOST, Assistant Professor, Ondokuz Mayıs University
Organization: Ondokuz Mayıs University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ESP0255
Record Dates: First submitted 2020-04-03; First posted 2020-04-07 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Prostate Cancer; Anesthesia, Local; Pain, Postoperative
Keywords: Pain, Postoperative; Ultrasound Guided Erector Spinae Plane Block; Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms; Pain, Postoperative | interventions — Parapsychology; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group LB (Active Comparator): Ultrasound-guided bilateral erector spinae plane block (10 ml 1% lidocaine + 10 ml 0.5% bupivacaine) + intravenous morphine patient-controlled analgesia.
  Interventions: Procedure: Single-injection ultrasound-guided bilateral erector spinae plane block-Lidocaine/Bupivacaine; Other: Pain follow-up and monitorization
- Group S (Sham Comparator): Ultrasound-guided bilateral erector spinae plane block. block (20 ml Normal Saline) + intravenous morphine patient-controlled analgesia.
  Interventions: Procedure: Single-injection ultrasound-guided bilateral erector spinae plane (ESP) block-Sham; Other: Pain follow-up and monitorization

INTERVENTIONS:
Procedure: Single-injection ultrasound-guided bilateral erector spinae plane (ESP) block-Sham — With the patient in the sitting position, 20 ml normal saline will be administered between the T11 spinous process and the erector spinae muscles with the guidance of an ultrasound probe placed on a parasagittal plane.
  Intraoperative analgesia: after anesthesia induction, paracetamol 1 gr intravenous (IV)+ tenoxicam 20 mg IV + morphine 0.05 mg/kg IV (max 4 mg).
  Postoperative analgesia: IV morphine patient-controlled analgesia (PCA) of 0.5 mg/ml morphine (demand dose 1 mg; lockout interval 8 m; 6 mg/h limit).
  Other Names: ESP block-Sham
  Arms: Group S
Procedure: Single-injection ultrasound-guided bilateral erector spinae plane block-Lidocaine/Bupivacaine — With the patient in the sitting position, 10 ml 1% lidocaine + 10 ml 0.5% bupivacaine will be administered between the T11 spinous process and the erector spinae muscles with the guidance of an ultrasound probe placed on a parasagittal plane.
  Intraoperative analgesia: After anesthesia induction, paracetamol 1 gr IV + tenoxicam 20 mg IV + morphine 0.05 mg/kg IV (max 4 mg).
  Postoperative analgesia: IV PCA of 0.5 mg/ml morphine (demand dose 1 mg; lockout interval 8 m; 6 mg/h limit).
  Other Names: ESP block-Lidocaine/Bupivacaine
  Arms: Group LB
Other: Pain follow-up and monitorization — Numeric Rating Scale (NRS) pain score will be recorded from 15th minute in recovery room followed by 1.-3.-6.-12.-18.-24.hours with two different conditions which are at rest and while couching.If NRS score becomes ≥4 Dexketoprofen 50 mg will be administered (max 4 times).
  Other Names: IV morphine-PCA

SUMMARY:
In the proposed study, a bilateral erector spinae plane (ESP) block [10 ml 1%lidocaine + 10 ml 0.5 % bupivacaine vs normal saline (NS)] will be performed preoperatively to patients undergoing open radical prostatectomy. Analgesic efficacy will be assessed on the numeric rating scale (NRS) along with intra- and 24 h post-operative narcotic consumption.

DETAILED DESCRIPTION:
It has been reported that the ESP block produces effective postoperative analgesia for abdominal surgeries by relieving both somatic and visceral pain. In the present study, the investigators presume that an ESP block will decrease narcotic consumption and NRS values both intraoperatively and during the first 24 postoperative hours.

Patients will be divided into two groups:

Group LB (Lidocaine-Bupivacaine): A bilateral ESP block will be performed preoperatively (10 ml 1%lidocaine + 10 ml 0.5% bupivacaine). In addition, IV morphine patient-controlled analgesia (PCA) will be applied postoperatively for 24 hours.

Group S: A bilateral ESP block will be performed preoperatively (20 ml NS).In addition, IV morphine-PCA will be applied postoperatively for 24 hours.

ELIGIBILITY:
Inclusion Criteria: AmericanSociety of Anesthesiologists (ASA) I-III patients between the ages of 18 and 65 who are scheduled for elective open radical prostatectomy.

Exclusion criteria:

* Patients who do not give informed consent or do not want to participate in the study
* Ages <18 or>65
* ASA IV patients
* Obesity (>100 kg, BMI >35 kg/m2)
* Contraindications of regional anesthesia (coagulopathy, thrombocytopenia, or infection at injection site)
* Serious renal, cardiac, or hepatic disease
* Hypersensitivity to local anesthetics or a history of allergy
* History of opioid or steroid use longer than four weeks
* Psychiatric disorders
* Analgesic preoperative treatment within the preceding 48 hours
* In order to establish better standard surgery, operations shorter than 60 minutes and longer than 180 minutes will also be excluded

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only Male
Enrollment: 52 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2021-01-11 (Actual)

PRIMARY OUTCOMES:
Narcotic consumption in the first 24 hours after surgery | Postoperative day 1
  Morphine consumption in the first 24 hours will be measured by IV PCA. Patients will be able to request opioids via a PCA device when their NRS score is above 3.

SECONDARY OUTCOMES:
Postoperative pain: NRS score | Postoperative day 1
  Pain status at rest and while coughing will be assessed by NRS score at 1, 3, 6, 12, 18, and 24 hours after surgery. In addition, the time until first analgesic requirement will be recorded.The NRS is an 11-point numeric scale which ranges from 0 to 10.
Postoperative nausea and vomiting (PONV) | Postoperative day 1
  The patients will be verbally evaluated according to a descriptive five-point PONV scale. If a score of 3 or more is registered, ondansetron 4 mg IV will be administered and repeated after 8 hours if required.The PONV scale is 0 = no nausea; 1 = slight nausea; 2 = moderate nausea; 3 = vomiting once;and 4 = vomiting more than once
Intraoperative remifentanil consumption | Postoperative day 1
  Following anesthesia induction, a bispectral index (BIS) of 40 to 50 will be maintained with sevoflurane. When the BIS measures 40-50, the remifentanil infusion rate will be adjusted to consider ±20% blood pressure changes compared to baseline values.The total amount of remifentanil consumed will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: BURHAN DOST, Study Director — Ondokuz Mayis University, School of Medicine, Department of Anesthesiology
Locations (1):
- Ondokuz Mayis University, Samsun, Atakum, Turkey (Türkiye)

REFERENCES:
- [Background] Ibrahim M, Elnabtity AM. Analgesic efficacy of erector spinae plane block in percutaneous nephrolithotomy : A randomized controlled trial. Anaesthesist. 2019 Nov;68(11):755-761. doi: 10.1007/s00101-019-00673-w. Epub 2019 Oct 16. PMID 31620856
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Chin KJ, Adhikary S, Sarwani N, Forero M. The analgesic efficacy of pre-operative bilateral erector spinae plane (ESP) blocks in patients having ventral hernia repair. Anaesthesia. 2017 Apr;72(4):452-460. doi: 10.1111/anae.13814. Epub 2017 Feb 11. PMID 28188621
- [Background] Diwan S, Nair A. Is Paravertebral-Epidural Spread the Underlying Mechanism of Action of Erector Spinae Plane Block? Turk J Anaesthesiol Reanim. 2020 Feb;48(1):86-87. doi: 10.5152/TJAR.2019.81226. Epub 2019 Nov 11. No abstract available. PMID 32076689
- [Background] Kot P, Rodriguez P, Granell M, Cano B, Rovira L, Morales J, Broseta A, Andres J. The erector spinae plane block: a narrative review. Korean J Anesthesiol. 2019 Jun;72(3):209-220. doi: 10.4097/kja.d.19.00012. Epub 2019 Mar 19. PMID 30886130
- [Background] Tulgar S, Kapakli MS, Kose HC, Senturk O, Selvi O, Serifsoy TE, Thomas DT, Ozer Z. Evaluation of Ultrasound-Guided Erector Spinae Plane Block and Oblique Subcostal Transversus Abdominis Plane Block in Laparoscopic Cholecystectomy: Randomized, Controlled, Prospective Study. Anesth Essays Res. 2019 Jan-Mar;13(1):50-56. doi: 10.4103/aer.AER_194_18. PMID 31031480 (Retraction: PMID 34092875 Anesth Essays Res. 2020 Jul-Sep;14(3):544)
- [Background] Singh S, Kumar G, Akhileshwar. Ultrasound-guided erector spinae plane block for postoperative analgesia in modified radical mastectomy: A randomised control study. Indian J Anaesth. 2019 Mar;63(3):200-204. doi: 10.4103/ija.IJA_758_18. PMID 30988534